CLINICAL TRIAL: NCT06466122
Title: Phase 2 Study of Combination Pirtobrutinib (LOXO-305) and Venetoclax in CLL Patients With Resistance to Covalent BTKi
Brief Title: Pirtobrutinib (LOXO-305) and Venetoclax for the Treatment of Patients With CLL or SLL Resistant to Covalent BTKi
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kerry Rogers (Other)
Responsible Party: Sponsor-Investigator, Kerry Rogers, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-22172; NCI-2024-04627 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-06-07; First posted 2024-06-20 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Specimen Handling; Biopsy; pirtobrutinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pirtobrutinib, venetoclax) (Experimental): Patients receive pirtobrutinib PO QD on days 1-28 of each cycle and receive venetoclax PO QD on days 1-28 of cycles 2-20. Cycles repeat every 28 days for up to 20 cycles in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression within 12 months of stopping combination treatment may receive pirtobrutinib PO QD in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy and CT throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Pirtobrutinib; Drug: Venetoclax

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Pirtobrutinib — Given PO
  Other Names: 5-Amino-3-(4-((5-fluoro-2-methoxybenzamido)methyl)phenyl)-1-((2S)-1,1,1-trifluoropropan-2-yl)-1h-pyrazole-4-carboxamide; BTK Inhibitor LOXO-305; Jaypirca; LOXO 305; LOXO-305; LOXO305; LY3527727
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial tests how well pirtobrutinib (LOXO-305) and venetoclax works in treating patients with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) that remains despite treatment (resistant) with covalent bruton tyrosine kinase inhibitors (BTKi). Pirtobrutinib is in a class of medications called kinase inhibitors. It works by blocking the action of the a protein that signals cancer cells to multiply. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking BCL-2, a protein needed for cancer cell survival. Giving pirtobrutinib and venetoclax may kill more cancer cells in patients with CLL or SLL that is resistant to covalent BTKi.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine if combination pirtobrutinib and venetoclax can induce undetectable minimal residual disease (uMRD) in CLL patients with resistance to ibrutinib, acalabrutinib, or zanubrutinib.

OUTLINE:

Patients receive pirtobrutinib orally (PO) once daily (QD) on days 1-28 of each cycle and receive venetoclax PO QD on days 1-28 of cycles 2-20. Cycles repeat every 28 days for up to 20 cycles in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression within 12 months of stopping combination treatment may receive pirtobrutinib PO QD in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, bone marrow aspiration and biopsy and computed tomography (CT) throughout the study.

After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL or SLL according to the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 guidelines
* Detectable CLL on flow cytometry of the blood or marrow at time of enrollment
* Age ≥ 18 years old
* Eastern Cooperative Oncology Group (ECOG) performance 0-2
* Currently taking ibrutinib, acalabrutinib, or zanubrutinib at any daily dose and tolerating it for > 4 weeks
* Evidence of progressive disease by iwCLL 2018 criteria for progressive disease or doubling of absolute lymphocyte count (ALC) in ≤ 6 months while on BTK inhibitor provided ALC is > 5 k/uL
* Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) ≤ 3 x the upper limit of normal (ULN) or ≤ 5 x ULN with documented liver involvement
* Bilirubin ≤ 1.5 x ULN or ≤ 3 x ULN with documented liver involvement and/or Gilbert's disease
* Creatinine clearance (CrCl) ≥ 30 according to modified Cockcroft-Gault equation
* Absolute neutrophil count (ANC) ≥ 0.75 k/uL

  * Without transfusion or growth factor administration in the 7 days prior to screening
  * Any values if cytopenias are due to bone marrow involvement with disease
* Hemoglobin ≥ 8 g/dL

  * Without transfusion or growth factor administration in the 7 days prior to screening
  * Any values if cytopenias are due to bone marrow involvement with disease
* Platelets ≥ 50 k/uL

  * Without transfusion or growth factor administration in the 7 days prior to screening
  * Any values if cytopenias are due to bone marrow involvement with disease
* Prothrombin time (PT) and partial thromboplastin time (PTT) ≤ 1.5 x ULN
* No known inherited qualitative platelet defect (e.g. delta granule storage pool deficiency)
* Willing and able to complete study activities and treatment
* Willing and capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol
* Willingness of men and women of reproductive potential and their partners to observe conventional and highly effective or acceptable birth control methods for the duration of treatment and for 6 months following the last dose of pirtobrutinib or 30 days from the last dose of venetoclax
* ELIGIBILITY FOR RE-TREATMENT WITH PIRTOBRUTINIB: Discontinued initial study treatment ≤ 12 months ago
* ELIGIBILITY FOR RE-TREATMENT WITH PIRTOBRUTINIB: Meets iwCLL 2018 criteria for progressive disease

Exclusion Criteria:

* Inability to tolerate 2 Liters of oral or intravenous (IV) hydration
* Prior venetoclax exposure > 13 months or known resistance to venetoclax
* Known hypersensitivity to any of the excipients of pirtobrutinib or venetoclax
* Need for treatment with warfarin or other vitamin K antagonist during study treatment
* History of bleeding diathesis
* Patients who experienced a major bleeding event or grade ≥ 3 arrhythmia on prior treatment with a BTK inhibitor. Major bleeding is defined as bleeding having one or more of the following features: potentially life-threatening bleeding with signs or symptoms of hemodynamic compromise; bleeding associated with a decrease in the hemoglobin level of at least 2g per deciliter; or bleeding in a critical area or organ (e.g., retroperitoneal, intraarticular, pericardial, epidural, or intracranial bleeding or intramuscular bleeding with compartment syndrome)
* History of stroke or intracranial hemorrhage within 6 months
* Inability to take pills or oral medications
* Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal (GI) absorption of either pirtobrutinib or venetoclax
* Current known central nervous system involvement with CLL or SLL. Patients with previous treatment for central nervous system (CNS) involvement who are neurologically stable and without evidence of disease may be eligible if a compelling clinical rationale is provided by the investigator and with documented approval by the principal investigator
* Treatment with the following:

  * Targeted agents, investigational agents, therapeutic monoclonal antibodies, or cytotoxic chemotherapy within 5 half-lives or 2 weeks, whichever is shorter
  * Treatment with immunoconjugated antibody treatment within 10 weeks
  * Receipt of broad field radiation ( ≥ 30% of the bone marrow or whole brain radiotherapy) within 14 days or palliative limited field radiation within 7 days prior to study enrollment
  * Note: Treatment with ibrutinib, acalabrutinib, or zanubrutinib is allowed. Treatment with topical chemotherapy agents for precancerous skin conditions or skin cancers is allowed
* Unresolved adverse events from prior treatment not resolved to grade ≤ 1 with the exception of alopecia or grade 2 peripheral neuropathy
* History of allogeneic or autologous stem cell transplant (SCT) or chimeric antigen receptor-modified T cell (CAR-T) therapy within 60 days. Patients with a history of allogeneic stem cell transplant must be stable off all immunosuppression for at least 2 months prior to study screening. Presence of any of the following, regardless of prior SCT and/or CAR-T therapy timing will be exclusionary:

  * Active graft versus host disease (GVHD)
  * Cytopenia from incomplete blood cell count recovery post-transplant
  * Need for anti-cytokine therapy for toxicity from CAR-T therapy and/or residual symptoms of neurotoxicity > grade 1 from CAR-T therapy
  * Ongoing immunosuppressive therapy
* Active second malignancy unless in remission and with life expectancy > 2 years. Adjuvant endocrine therapy for breast or prostate cancer that is expected to be cured is allowed. Non-melanoma skin cancers are permitted if adequately treated
* Psychiatric illness, or social situations that would limit compliance with study requirements
* Active uncontrolled auto-immune cytopenia (e.g., autoimmune hemolytic anemia [AIHA], idiopathic thrombocytopenic purpura [ITP]) for which new therapy was introduced or existing therapy was escalated within the 4 weeks prior to study enrollment to maintain adequate blood counts
* Evidence of other clinically significant uncontrolled condition(s) including but not limited to, uncontrolled systemic bacterial, viral, fungal or parasitic infection (except for fungal nail infection), or other clinically significant active disease process which in the opinion of the investigator may pose a risk for patient participation. Screening for chronic conditions is not required
* Significant cardiovascular disease defined as:

  * Unstable angina or acute coronary syndrome within the past 2 months
  * History of myocardial infarction within 3 months
  * Documented left ventricular ejection fraction (LVEF) by any method of ≤ 40% in the 12 months
  * ≥ grade 3 New York Heart Association (NYHA) functional classification system of heart failure
  * Uncontrolled or symptomatic arrhythmias
* Prolongation of the QT interval corrected for heart rate (Fridericia's formula-corrected QT interval [QTcF]) > 470 msec. QTcF is calculated using Fridericia's formula

  * Correction of suspected drug induced QTcF prolongation can be attempted at the investigator¡¦s discretion and only if clinically safe to do so with either discontinuation of the offending drug or switch to another drug not known to be associated with QTcF prolongation
  * Correction for underlying bundle branch block (BBB) allowed
  * Note: Patients with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection based on criteria below:

  * Hepatitis B virus (HBV): Patients with positive hepatitis B surface antigen (HBsAg) are excluded. Patients with positive hepatitis B core antibody (anti-HBc) and negative HBsAg require hepatitis B polymerase chain reaction (PCR) evaluation before inclusion. Patients who are hepatitis B PCR positive will be excluded
  * Hepatitis C virus (HCV): positive hepatitis C antibody. If positive hepatitis C antibody result, patient will need to have a negative result for hepatitis C ribonucleic acid (RNA) before inclusion. Patients who are hepatitis C RNA positive will be excluded. Patients previously treated for hepatitis C > 6 months previously with a negative RNA test are eligible
* Known HIV infection. For patients with unknown HIV status, HIV testing will be performed at screening and result should be negative for enrollment
* Known active cytomegalovirus (CMV) infection. Unknown or negative status are eligible
* Treatment with a strong CYP3A inhibitor or inducer and/or strong P-gp inhibitors within 3 days of starting or during study treatment. Treatment with a moderate or strong CYP3A inhibitor or inducer within 7 days prior to first dose of venetoclax or during cycle 2 or 3 of study treatment. Patients may not plan to consume grapefruit or grapefruit products, Seville oranges or products from Seville oranges, or star fruit
* Pregnancy, lactation, or plan to breastfeed during the study or within 6 months of the last dose of either pirtobrutinib or venetoclax
* Major surgery within 4 weeks prior to screening
* Vaccination with live vaccine within 28 days of screening
* Currently incarcerated
* History of progressive multifocal leukoencephalopathy (PML) or human polyomavirus 2 (JC virus) infection
* History of seizure disorder unless controlled without a seizure in the year prior to screening
* ELIGIBILITY FOR RE-TREATMENT WITH PIRTOBRUTINIB: Has not developed any new medical conditions that would change the safety of treatment with pirtobrutinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of undetectable minimal residual disease (uMRD) | At cycle 21 day 1 (C21D1) [each cycle lasts 28 days]
  The rate of uMRD will be defined as the percentage of patients who have uMRD in both the peripheral blood and bone marrow at C21D1.

SECONDARY OUTCOMES:
Best overall response rate (ORR) | At cycle 21 day 1 (C21D1) [each cycle lasts 28 days]
  Best ORR will be estimated with exact 95% confidence intervals.
Overall Response Rate (ORR) | At cycle 21 day 1 (C21D1) [each cycle lasts 28 days]
  ORR will be estimated with exact 95% confidence intervals.
Progression-free survival (PFS) for all patients | At start of treatment to progression or death up to 18 months after completion of study treatment
  Clinical disease progression will be assessed by International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 criteria. PFS will be described using the method of Kaplan-Meier. Median and/or estimates at clinically meaningful time points for PFS will be reported with 95% confidence intervals.
PFS in patients who achieve uMRD and those who do not achieve uMRD with pirtobrutinib and venetoclax | At end of treatment to progression or death up to 18 months after completion of study treatment
  Clinical disease progression will be assessed by iwCLL 2018 criteria. PFS will be described using the method of Kaplan-Meier. Median and/or estimates at clinically meaningful time points for PFS will be reported with 95% confidence intervals.
Overall survival (OS) for all patients | At start of treatment to death up to 18 months after completion of study treatment
  OS will be described using the method of Kaplan-Meier. Median and/or estimates at clinically meaningful time points for OS will be reported with 95% confidence intervals.
OS for patients who achieve uMRD and those who do not achieve uMRD with pirtobrutinib and venetoclax | At end of treatment to death up to 18 months after completion of study treatment
  OS will be described using the method of Kaplan-Meier. Median and/or estimates at clinically meaningful time points for OS will be reported with 95% confidence intervals.
Incidence of adverse events (AEs) | Up to 28 days after last dose of study drugs
  AEs will be summarized by type, severity and perceived attribution according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Hematologic AEs will be graded according to CLL specific criteria described in the iwCLL 2018 guidelines. The maximum grade for each type of AE will be recorded for each patient, and at a minimum, frequency tables will be reviewed to determine AE patterns. The number of patients who discontinue treatment due to AE will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Kerry A Rogers, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu